CLINICAL TRIAL: NCT03068793
Title: Multimodal Neural Investigation of Reward Processing in Mental Illness
Brief Title: Reward Processing in Mental Illness
Status: Completed | Type: Observational
Sponsor: Susanna Fryer (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Susanna Fryer, Assistant Professor in Residence, San Francisco Veterans Affairs Medical Center
Organization: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Other Study IDs: IK2CX001028 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Early-onset Schizophrenia
MeSH Terms: interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with Recent Onset Schizophrenia: Individuals who have been diagnosed with Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder within the past five years and meet our research criteria for symptoms indicative of these diseases within the past five years.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Patients with Major Depressive Disorder: Individuals who have been diagnosed with Major Depressive Disorder within the past five years and meet our research criteria for symptoms indicative of this disease within the past five years.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Patients with Gambling Disorder: Individuals who have been diagnosed with Gambling Disorder within the past five years and meet our research criteria for symptoms indicative of this disease within the past five years.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Patients with Post Traumatic Stress Disorder: Individuals who have been diagnosed with Post Traumatic Stress Disorder within the past five years and meet our research criteria for symptoms indicative of this disease within the past five years.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)
- Healthy Controls: Individuals who have not met criteria for a psychiatric, mood, or gambling disorder within their lifetime according to our research criteria for symptoms indicative of a psychiatric, mood, or gambling disorder.
  Interventions: Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Electroencephalography (EEG) and Magnetic Resonance Imaging (MRI) — We will use these techniques combined with tests of reward anticipation and clinical interviews to explore connections between these measures and activity in the brain in patients with a diagnosis of schizophrenia, major depressive disorder, gambling disorder, or post traumatic stress disorder and healthy controls.

SUMMARY:
The purpose of this study is to examine the nature of reward processing dysfunctions in schizophrenia using neuroimaging techniques that capture in vivo brain functioning, such as EEG and fMRI.

DETAILED DESCRIPTION:
This experiment takes place over the course of two or three days. On each visit day, the experiment will involve a brief interview session, electroencephalography (EEG) recording,and/or a magnetic resonance imaging (MRI).

Screening tests or procedures include:

* If you are female of child bearing potential, you must complete a urine pregnancy test for the MRI procedure
* You will be asked a series of questions about your mental health and your background

If the screening exam shows that you can be in the main part of the study and you choose to continue, these are the tests and procedures that you would complete on one or two test days:

* EEG recording: In this procedure, the researcher will assess your brain function while you perform simple computer-based tasks. The computer tasks involve presentation of pictures to which you respond by pressing a button. You will be given clear instructions and a chance to practice before each task. While you are performing these tasks, we will record the weak electrical signals produced by your brain, or "brain waves", using a technique called electroencephalography (EEG).

  * In order to record your EEG, sensors (small plastic discs) will be attached to specific locations on your scalp. Your scalp will be gently scrubbed before the sensors are attached. The sensors are held in place on your scalp using a nylon cap that fits snugly on your head. Sensors will also be attached above and below your eyes and will record your eye movements. It will take approximately one hour to attach the sensors. The entire EEG will take approximately 2 hours.
  * Before you take part in the EEG session, please make sure to wash your hair and scalp. Do not use conditioner or a 2-in-1 shampoo/conditioner. Your hair should be dry before your arrival. We ask this in order to make the set-up process go more smoothly.
* MRI: In the fMRI procedure, we will use a magnet to measure blood flow to your brain while you do different cognitive tasks. You will be asked to lie down on a platform that can be slid into the middle of the magnet. A plastic MRI imaging coil will be placed around your head. You will not come into contact with the coil during the experiment. Foam pads will be placed around your head to limit head movement during the experiment. We will then slide you into the magnet. At different points during the experiment, you will be asked to do the same tasks you did in the training session prior to the scan. During the scan, you will be asked to either lie still and rest, or do some tasks similar to those you completed during your EEG. The entire MRI will take approximately two hours.

  * If the researchers feel as though the quality of data collected by the scanner can be improved, you may be asked to return for an additional scan session.
* Brief interview session: There will be a series of questions about your education, smoking status, and economic background. You will also be given a list of words to read to the researcher. If you are a patient diagnosed with one of the above-mentioned psychiatric disorders, you will be asked to participate in an additional interview, lasting about one hour, focusing on how you have been feeling recently.

ELIGIBILITY:
Inclusion Criteria:

* The subject population will include 18 to 30 year old participants of any gender, race, and ethnicity. All subjects will be able to speak and understand English.

Schizophrenia subjects:

1. Patients must be diagnosed with DSM-IV schizophrenia, schizophreniform, or schizoaffective disorder based on a SCID-P interview.

Depression subjects:

1. Patients must be diagnosed with DSM-V Major Depressive Disorder based on a SCID-P interview.

Post Traumatic Stress Disorder subjects:

1. Patients must be diagnosed with DSM-V Post Traumatic Stress Disorder based on a SCID-P interview.

Gambling Disorder subjects:

1. Patients must be diagnosed with DSM-V Gambling Disorder based on a SCID-P interview.

Comparison subjects:

1. Control participants must not have past or present Axis I diagnosis as determined by the SCID-NP.

Exclusion Criteria:

* All subjects:

  1. A hearing deficit greater than 40dB in both ears detected during the hearing test
  2. Substance dependence, as per clinical judgment, in the past 1 year (except caffeine and nicotine)
  3. A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic or neurological
  4. History of head injury with loss of consciousness greater than 15 minutes
  5. Any other condition or medication, which in the opinion of the investigator would preclude participation in the study.
  6. Non-English speaking.

Comparison subjects:

1. Any first-degree relative with schizophrenia or bipolar disorder.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have been diagnosed with schizophrenia, schizoaffective disorder, or schizophreniform disorder within the past 5 years and meet our research criteria of symptoms indicative of a diagnosis of schizophrenia within their lifetime are eligible for this study.
  Patients who have been diagnosed with Major Depressive Disorder, Post Traumatic Stress Disorder, and Gambling Disorder within the past 5 years and meet our research criteria of symptoms indicative of a diagnosis of one of these disorders within their lifetime are also eligible for this study.
  Healthy controls who have never met criteria for a psychiatric disorder and meet our research criteria will also be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
EEG | At time of visit
  Electroencephalography, measures signals from the brain while participants conduct specific tasks that measure memory and attention.
MRI | At time of visit
  Magnetic Resonance Imaging, measures activity in, and takes detailed pictures of the brain while participants conduct specific tasks that measure memory and attention.
Reward Processing Tasks | At time of visit
  A slot machine task where participants can win real money while participating in an EEG and MRI

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Fryer, PhD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fenton WS, McGlashan TH. Natural history of schizophrenia subtypes. II. Positive and negative symptoms and long-term course. Arch Gen Psychiatry. 1991 Nov;48(11):978-86. doi: 10.1001/archpsyc.1991.01810350018003. PMID 1747021
- [Background] Bleuler, E. Dementia Praecox or the Group of Schizophrenias. (1911) (International Universities Press, New York, NY, Translated by J. Zinkin, 1950).
- [Background] Milev P, Ho BC, Arndt S, Andreasen NC. Predictive values of neurocognition and negative symptoms on functional outcome in schizophrenia: a longitudinal first-episode study with 7-year follow-up. Am J Psychiatry. 2005 Mar;162(3):495-506. doi: 10.1176/appi.ajp.162.3.495. PMID 15741466
- [Background] Rabinowitz J, Levine SZ, Garibaldi G, Bugarski-Kirola D, Berardo CG, Kapur S. Negative symptoms have greater impact on functioning than positive symptoms in schizophrenia: analysis of CATIE data. Schizophr Res. 2012 May;137(1-3):147-50. doi: 10.1016/j.schres.2012.01.015. Epub 2012 Feb 6. PMID 22316568
- [Background] Kirkpatrick B, Fenton WS, Carpenter WT Jr, Marder SR. The NIMH-MATRICS consensus statement on negative symptoms. Schizophr Bull. 2006 Apr;32(2):214-9. doi: 10.1093/schbul/sbj053. Epub 2006 Feb 15. No abstract available. PMID 16481659
- [Background] Gold JM, Waltz JA, Matveeva TM, Kasanova Z, Strauss GP, Herbener ES, Collins AG, Frank MJ. Negative symptoms and the failure to represent the expected reward value of actions: behavioral and computational modeling evidence. Arch Gen Psychiatry. 2012 Feb;69(2):129-38. doi: 10.1001/archgenpsychiatry.2011.1269. PMID 22310503
- [Background] Gold JM, Waltz JA, Prentice KJ, Morris SE, Heerey EA. Reward processing in schizophrenia: a deficit in the representation of value. Schizophr Bull. 2008 Sep;34(5):835-47. doi: 10.1093/schbul/sbn068. Epub 2008 Jun 30. PMID 18591195
- [Background] Heinz A, Schlagenhauf F. Dopaminergic dysfunction in schizophrenia: salience attribution revisited. Schizophr Bull. 2010 May;36(3):472-85. doi: 10.1093/schbul/sbq031. Epub 2010 May 7. PMID 20453041
- [Background] Waltz JA, Frank MJ, Robinson BM, Gold JM. Selective reinforcement learning deficits in schizophrenia support predictions from computational models of striatal-cortical dysfunction. Biol Psychiatry. 2007 Oct 1;62(7):756-64. doi: 10.1016/j.biopsych.2006.09.042. Epub 2007 Feb 14. PMID 17300757
- [Background] Barch DM, Dowd EC. Goal representations and motivational drive in schizophrenia: the role of prefrontal-striatal interactions. Schizophr Bull. 2010 Sep;36(5):919-34. doi: 10.1093/schbul/sbq068. Epub 2010 Jun 21. PMID 20566491
- [Background] Haber SN, Knutson B. The reward circuit: linking primate anatomy and human imaging. Neuropsychopharmacology. 2010 Jan;35(1):4-26. doi: 10.1038/npp.2009.129. PMID 19812543
- [Background] Maldjian JA, Laurienti PJ, Kraft RA, Burdette JH. An automated method for neuroanatomic and cytoarchitectonic atlas-based interrogation of fMRI data sets. Neuroimage. 2003 Jul;19(3):1233-9. doi: 10.1016/s1053-8119(03)00169-1. PMID 12880848
- [Background] Schultz W. Behavioral theories and the neurophysiology of reward. Annu Rev Psychol. 2006;57:87-115. doi: 10.1146/annurev.psych.56.091103.070229. PMID 16318590
- [Background] Schultz W, Dayan P, Montague PR. A neural substrate of prediction and reward. Science. 1997 Mar 14;275(5306):1593-9. doi: 10.1126/science.275.5306.1593. PMID 9054347
- [Background] Berridge KC. The debate over dopamine's role in reward: the case for incentive salience. Psychopharmacology (Berl). 2007 Apr;191(3):391-431. doi: 10.1007/s00213-006-0578-x. Epub 2006 Oct 27. PMID 17072591
- [Background] Miller R. Schizophrenic psychology, associative learning and the role of forebrain dopamine. Med Hypotheses. 1976 Sep-Oct;2(5):203-11. doi: 10.1016/0306-9877(76)90040-2. PMID 9558
- [Background] Stein L, Wise CD. Possible etiology of schizophrenia: progressive damage to the noradrenergic reward system by 6-hydroxydopamine. Science. 1971 Mar 12;171(3975):1032-6. doi: 10.1126/science.171.3975.1032. PMID 5100789
- [Background] Kapur S. Psychosis as a state of aberrant salience: a framework linking biology, phenomenology, and pharmacology in schizophrenia. Am J Psychiatry. 2003 Jan;160(1):13-23. doi: 10.1176/appi.ajp.160.1.13. PMID 12505794
- [Background] Bromberg-Martin ES, Matsumoto M, Hikosaka O. Dopamine in motivational control: rewarding, aversive, and alerting. Neuron. 2010 Dec 9;68(5):815-34. doi: 10.1016/j.neuron.2010.11.022. PMID 21144997
- [Background] Esslinger C, Englisch S, Inta D, Rausch F, Schirmbeck F, Mier D, Kirsch P, Meyer-Lindenberg A, Zink M. Ventral striatal activation during attribution of stimulus saliency and reward anticipation is correlated in unmedicated first episode schizophrenia patients. Schizophr Res. 2012 Sep;140(1-3):114-21. doi: 10.1016/j.schres.2012.06.025. Epub 2012 Jul 10. PMID 22784688
- [Background] Juckel G, Schlagenhauf F, Koslowski M, Wustenberg T, Villringer A, Knutson B, Wrase J, Heinz A. Dysfunction of ventral striatal reward prediction in schizophrenia. Neuroimage. 2006 Jan 15;29(2):409-16. doi: 10.1016/j.neuroimage.2005.07.051. Epub 2005 Sep 1. PMID 16139525
- [Background] Nielsen MO, Rostrup E, Wulff S, Bak N, Lublin H, Kapur S, Glenthoj B. Alterations of the brain reward system in antipsychotic naive schizophrenia patients. Biol Psychiatry. 2012 May 15;71(10):898-905. doi: 10.1016/j.biopsych.2012.02.007. Epub 2012 Mar 13. PMID 22418013
- [Background] Schlagenhauf F, Juckel G, Koslowski M, Kahnt T, Knutson B, Dembler T, Kienast T, Gallinat J, Wrase J, Heinz A. Reward system activation in schizophrenic patients switched from typical neuroleptics to olanzapine. Psychopharmacology (Berl). 2008 Mar;196(4):673-84. doi: 10.1007/s00213-007-1016-4. Epub 2007 Dec 21. PMID 18097655
- [Background] Schlagenhauf F, Sterzer P, Schmack K, Ballmaier M, Rapp M, Wrase J, Juckel G, Gallinat J, Heinz A. Reward feedback alterations in unmedicated schizophrenia patients: relevance for delusions. Biol Psychiatry. 2009 Jun 15;65(12):1032-9. doi: 10.1016/j.biopsych.2008.12.016. Epub 2009 Feb 5. PMID 19195646
- [Background] Dowd EC, Barch DM. Pavlovian reward prediction and receipt in schizophrenia: relationship to anhedonia. PLoS One. 2012;7(5):e35622. doi: 10.1371/journal.pone.0035622. Epub 2012 May 4. PMID 22574121
- [Background] Simon JJ, Biller A, Walther S, Roesch-Ely D, Stippich C, Weisbrod M, Kaiser S. Neural correlates of reward processing in schizophrenia--relationship to apathy and depression. Schizophr Res. 2010 May;118(1-3):154-61. doi: 10.1016/j.schres.2009.11.007. Epub 2009 Dec 16. PMID 20005675
- [Background] Waltz JA, Schweitzer JB, Ross TJ, Kurup PK, Salmeron BJ, Rose EJ, Gold JM, Stein EA. Abnormal responses to monetary outcomes in cortex, but not in the basal ganglia, in schizophrenia. Neuropsychopharmacology. 2010 Nov;35(12):2427-39. doi: 10.1038/npp.2010.126. Epub 2010 Aug 18. PMID 20720534
- [Background] Knutson B, Adams CM, Fong GW, Hommer D. Anticipation of increasing monetary reward selectively recruits nucleus accumbens. J Neurosci. 2001 Aug 15;21(16):RC159. doi: 10.1523/JNEUROSCI.21-16-j0002.2001. PMID 11459880
- [Background] Gard DE, Kring AM, Gard MG, Horan WP, Green MF. Anhedonia in schizophrenia: distinctions between anticipatory and consummatory pleasure. Schizophr Res. 2007 Jul;93(1-3):253-60. doi: 10.1016/j.schres.2007.03.008. Epub 2007 May 9. PMID 17490858
- [Background] Horan WP, Wynn JK, Kring AM, Simons RF, Green MF. Electrophysiological correlates of emotional responding in schizophrenia. J Abnorm Psychol. 2010 Feb;119(1):18-30. doi: 10.1037/a0017510. PMID 20141239
- [Background] Kring AM, Moran EK. Emotional response deficits in schizophrenia: insights from affective science. Schizophr Bull. 2008 Sep;34(5):819-34. doi: 10.1093/schbul/sbn071. Epub 2008 Jun 25. PMID 18579556
- [Background] Koch K, Schachtzabel C, Wagner G, Schikora J, Schultz C, Reichenbach JR, Sauer H, Schlosser RG. Altered activation in association with reward-related trial-and-error learning in patients with schizophrenia. Neuroimage. 2010 Mar;50(1):223-32. doi: 10.1016/j.neuroimage.2009.12.031. Epub 2009 Dec 16. PMID 20006717
- [Background] Morris RW, Vercammen A, Lenroot R, Moore L, Langton JM, Short B, Kulkarni J, Curtis J, O'Donnell M, Weickert CS, Weickert TW. Disambiguating ventral striatum fMRI-related BOLD signal during reward prediction in schizophrenia. Mol Psychiatry. 2012 Mar;17(3):235, 280-9. doi: 10.1038/mp.2011.75. Epub 2011 Jun 28. PMID 21709684
- [Background] Murray GK, Corlett PR, Clark L, Pessiglione M, Blackwell AD, Honey G, Jones PB, Bullmore ET, Robbins TW, Fletcher PC. Substantia nigra/ventral tegmental reward prediction error disruption in psychosis. Mol Psychiatry. 2008 Mar;13(3):239, 267-76. doi: 10.1038/sj.mp.4002058. Epub 2007 Aug 7. PMID 17684497
- [Background] Miltner WH, Braun CH, Coles MG. Event-related brain potentials following incorrect feedback in a time-estimation task: evidence for a "generic" neural system for error detection. J Cogn Neurosci. 1997 Nov;9(6):788-98. doi: 10.1162/jocn.1997.9.6.788. PMID 23964600
- [Background] Gehring WJ, Willoughby AR. The medial frontal cortex and the rapid processing of monetary gains and losses. Science. 2002 Mar 22;295(5563):2279-82. doi: 10.1126/science.1066893. PMID 11910116
- [Background] Walsh MM, Anderson JR. Learning from experience: event-related potential correlates of reward processing, neural adaptation, and behavioral choice. Neurosci Biobehav Rev. 2012 Sep;36(8):1870-84. doi: 10.1016/j.neubiorev.2012.05.008. Epub 2012 Jun 7. PMID 22683741
- [Background] Horan WP, Foti D, Hajcak G, Wynn JK, Green MF. Impaired neural response to internal but not external feedback in schizophrenia. Psychol Med. 2012 Aug;42(8):1637-47. doi: 10.1017/S0033291711002819. Epub 2011 Dec 8. PMID 22152069
- [Background] Morris SE, Holroyd CB, Mann-Wrobel MC, Gold JM. Dissociation of response and feedback negativity in schizophrenia: electrophysiological and computational evidence for a deficit in the representation of value. Front Hum Neurosci. 2011 Oct 28;5:123. doi: 10.3389/fnhum.2011.00123. eCollection 2011. PMID 22065618
- [Background] Morris SE, Heerey EA, Gold JM, Holroyd CB. Learning-related changes in brain activity following errors and performance feedback in schizophrenia. Schizophr Res. 2008 Feb;99(1-3):274-85. doi: 10.1016/j.schres.2007.08.027. Epub 2007 Sep 24. PMID 17889510
- [Background] Roiser JP, Stephan KE, den Ouden HE, Barnes TR, Friston KJ, Joyce EM. Do patients with schizophrenia exhibit aberrant salience? Psychol Med. 2009 Feb;39(2):199-209. doi: 10.1017/S0033291708003863. Epub 2008 Jun 30. PMID 18588739
- [Background] Chiew KS, Braver TS. Positive affect versus reward: emotional and motivational influences on cognitive control. Front Psychol. 2011 Oct 19;2:279. doi: 10.3389/fpsyg.2011.00279. eCollection 2011. PMID 22022318
- [Background] Pessoa L. How do emotion and motivation direct executive control? Trends Cogn Sci. 2009 Apr;13(4):160-6. doi: 10.1016/j.tics.2009.01.006. Epub 2009 Mar 13. PMID 19285913
- [Background] Savine AC, Braver TS. Motivated cognitive control: reward incentives modulate preparatory neural activity during task-switching. J Neurosci. 2010 Aug 4;30(31):10294-305. doi: 10.1523/JNEUROSCI.2052-10.2010. PMID 20685974 (Retraction: PMID 23678133 J Neurosci. 2013 May 15;33(20):8922)
- [Background] Locke HS, Braver TS. Motivational influences on cognitive control: behavior, brain activation, and individual differences. Cogn Affect Behav Neurosci. 2008 Mar;8(1):99-112. doi: 10.3758/cabn.8.1.99. PMID 18405050
- [Background] Small DM, Gitelman D, Simmons K, Bloise SM, Parrish T, Mesulam MM. Monetary incentives enhance processing in brain regions mediating top-down control of attention. Cereb Cortex. 2005 Dec;15(12):1855-65. doi: 10.1093/cercor/bhi063. Epub 2005 Mar 2. PMID 15746002
- [Background] Jimura K, Locke HS, Braver TS. Prefrontal cortex mediation of cognitive enhancement in rewarding motivational contexts. Proc Natl Acad Sci U S A. 2010 May 11;107(19):8871-6. doi: 10.1073/pnas.1002007107. Epub 2010 Apr 26. PMID 20421489
- [Background] Krawczyk DC, Gazzaley A, D'Esposito M. Reward modulation of prefrontal and visual association cortex during an incentive working memory task. Brain Res. 2007 Apr 13;1141:168-77. doi: 10.1016/j.brainres.2007.01.052. Epub 2007 Jan 25. PMID 17320835
- [Background] Taylor SF, Welsh RC, Wager TD, Phan KL, Fitzgerald KD, Gehring WJ. A functional neuroimaging study of motivation and executive function. Neuroimage. 2004 Mar;21(3):1045-54. doi: 10.1016/j.neuroimage.2003.10.032. PMID 15006672
- [Background] O'Connor DA, Rossiter S, Yucel M, Lubman DI, Hester R. Successful inhibitory control over an immediate reward is associated with attentional disengagement in visual processing areas. Neuroimage. 2012 Sep;62(3):1841-7. doi: 10.1016/j.neuroimage.2012.05.040. Epub 2012 May 25. PMID 22641143
- [Background] Egner T, Hirsch J. Cognitive control mechanisms resolve conflict through cortical amplification of task-relevant information. Nat Neurosci. 2005 Dec;8(12):1784-90. doi: 10.1038/nn1594. Epub 2005 Nov 6. PMID 16286928
- [Background] Watanabe M, Sakagami M. Integration of cognitive and motivational context information in the primate prefrontal cortex. Cereb Cortex. 2007 Sep;17 Suppl 1:i101-9. doi: 10.1093/cercor/bhm067. PMID 17725993
- [Background] Braver TS, Barch DM, Cohen JD. Cognition and control in schizophrenia: a computational model of dopamine and prefrontal function. Biol Psychiatry. 1999 Aug 1;46(3):312-28. doi: 10.1016/s0006-3223(99)00116-x. PMID 10435197
- [Background] Cohen JD, Braver TS, Brown JW. Computational perspectives on dopamine function in prefrontal cortex. Curr Opin Neurobiol. 2002 Apr;12(2):223-9. doi: 10.1016/s0959-4388(02)00314-8. PMID 12015241
- [Background] Fryer SL, Jorgensen KW, Yetter EJ, Daurignac EC, Watson TD, Shanbhag H, Krystal JH, Mathalon DH. Differential brain response to alcohol cue distractors across stages of alcohol dependence. Biol Psychol. 2013 Feb;92(2):282-91. doi: 10.1016/j.biopsycho.2012.10.004. Epub 2012 Nov 3. PMID 23131612
- [Background] Kriegeskorte N, Lindquist MA, Nichols TE, Poldrack RA, Vul E. Everything you never wanted to know about circular analysis, but were afraid to ask. J Cereb Blood Flow Metab. 2010 Sep;30(9):1551-7. doi: 10.1038/jcbfm.2010.86. Epub 2010 Jun 23. PMID 20571517
- [Background] First, M., Spitzer, R., Gibbon, M. & Williams, J. Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Patient Edition. (SCID-I/P). (New York State Psychiatric Institute, 2002).
- [Background] Horan WP, Kring AM, Gur RE, Reise SP, Blanchard JJ. Development and psychometric validation of the Clinical Assessment Interview for Negative Symptoms (CAINS). Schizophr Res. 2011 Nov;132(2-3):140-5. doi: 10.1016/j.schres.2011.06.030. Epub 2011 Jul 27. PMID 21798716
- [Background] Kring AM, Gur RE, Blanchard JJ, Horan WP, Reise SP. The Clinical Assessment Interview for Negative Symptoms (CAINS): final development and validation. Am J Psychiatry. 2013 Feb;170(2):165-72. doi: 10.1176/appi.ajp.2012.12010109. PMID 23377637
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Hollingshead AB, Redlich FC. Social class and mental illness: a community study. 1958. Am J Public Health. 2007 Oct;97(10):1756-7. doi: 10.2105/ajph.97.10.1756. No abstract available. PMID 17895405
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Fagerstrom KO. Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addict Behav. 1978;3(3-4):235-41. doi: 10.1016/0306-4603(78)90024-2. No abstract available. PMID 735910
- [Background] Wechsler, D. Wechsler Test of Adult Reading., (Psychological Corporation, 2001).
- [Background] Weissman, A. The Dysfunctional Attitudes Scale: A validation study., University of Pennsylvania, (1973).
- [Background] Carver, C. S. & White, T. L. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS Scales. Journal of Personality and Social Psychology 67,319-333 (1994).